CLINICAL TRIAL: NCT04883359
Title: Development of Immersive VR Environments to Induce and Evaluate Cognitive Fatigability: User Experience and Healthy Control Studies
Brief Title: Immersive VR Environments to Induce and Evaluate Cognitive Fatigability
Status: Terminated | Type: Observational
Why Stopped: PI left the NIH. Study will not continue.
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001744; 001744-NR
Record Dates: First submitted 2021-05-11; First posted 2021-05-12 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Cognitive Fatigue
Keywords: Emotional Regulation; Cognitive Interference; Planning; Behavioral Regulation; Stress Impact on Cognition; Natural History
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: From the Washington, D.C. metropolitan area

SUMMARY:
Background:

Immersive virtual reality (VR) technology is used by researchers to measure how people respond to complex stimuli in a controlled environment. Cognitive fatigue (CF) can result in serious consequences such as mistakes and accidents. Researchers want to see if VR can be used to learn more about CF.

Objective:

To test the user experience of a VR program designed to study individual differences in the susceptibility to develop CF in healthy people while performing activities of daily living.

Eligibility:

Healthy adults ages 18-75 from the Washington Metropolitan area

Design:

Participants will be screened with questions about their health and medical history.

The VR program simulates a real-world grocery shopping environment. Participants will be given a shopping task.

Participants will be seated. They will wear a head-mounted display (HMD) for 1.5 hours. The device is worn on the head. It presents images to the eyes. Eye-tracking data may be collected through the HMD.

The following will happen in the VR environment:

* Participants will be seated at a kitchen table. They will complete a pillbox task 2 times.
* Participants will be placed in a small grocery store. They will be trained how to use the controllers to shop.
* Participants will appear to be seated in front of a screen. They will be shown how to answer questions about how tired they feel and if the tasks are hard to do.
* Participants will be placed in a large grocery store. They will complete a shopping task.

Participants will complete surveys. They will also answer questions about the VR experience.

Participants will have 1 or 2 study visits. It will last 3-4 hours total.

DETAILED DESCRIPTION:
Objective: This study evaluates the utility of immersive virtual environments for objectively studying individual differences in the susceptibility to develop cognitive fatigue in healthy controls while performing instrumental activities of daily living (IADL) in two phases. Phase 1 aims to test functionality and user experience of the virtual reality (VR) experience; and phase 2 aims to evaluate the level of fatigue experienced after participating in a VR experience as measured by the Visual Analog Scale-Fatigue (VAS-F). The primary goal of the protocol is the study of individual differences in subjective fatigability associated with grocery shopping using immersive Virtual Reality as a research platform. The secondary objective of the protocol is to identify objective measures of cognitive fatigue.

Primary Endpoint Phase 1: The phase 1 primary dependent measure is the total count of the number of times, after completing the grocery shopping training exercise, the subject required research staff to explain how to use the controller, how to move or inspect objects, and/or how to move from one location to another location in the grocery store environment. Secondary Endpoint for Phase 1: the ocular and general symptoms score from the virtual reality symptom questionnaire (Ames et al., 2005); and the total score from the presence questionnaire (Regenbrecht et al., 2002).

The Primary Endpoint for Phase 2 primary:Total score of VAS-F (Lee et al., 1991).

The Secondary Endpoint for Phase 2;Self-reported cognitive load score measured by the NASA-TLX (Hart et al., 1988), eye-tracking data (e.g., percent eye-closure, fixation length, blink rate) and task performance measures (e.g. shopping list total correct item selection score, shopping list total incorrect item selection score, average item-selection time score).

Study Population: The study plans to enroll a total of 84 (24 in phase 1 and 60 in phase 2) healthy participants from the Washington Metropolitan area between ages 18-75.

Key Inclusion/Exclusion Criteria: Both study phases utilize the same key inclusion/exclusion. Participants must be between the ages (Bullet) 18 and 75 years. Key exclusion criteria include: visual impairment in the form of limited or reduced 3D vision, oculomotor disorder/dysfunction, susceptibility to visually-induced seizures, iritis, frequent headaches/migraines, severe sensitivity to motion sickness and any impairment in the use of arms/hands/fingers.

Design: All participants will complete the study at the NIH main campus clinical center. This is a two-phase research study. All participants will be screened for physical health, cognitive and visual symptoms via self-report. Phase 1 combines a traditional user experience design that utilizes qualitative, quantitative, and observational methods to test the software functionality, user interface, and realism of the immersive experience and a randomized control trial to estimate of effectiveness of the fatigue induction tasks. Phase 2 utilizes a 3-arm randomized control trial, where participants will be randomized into one of three virtual shopping experiences, a control condition (exploration of the shopping environment), a cognitively challenging condition (standard shopping list completion task), or a cognitive and emotionally challenging condition (shopping list with interruptions, interference, and rework). All participants will complete questionnaires and cognitive tests pre-and-post VR environment. Questionnaires related to target processes (fatigue and workload) are administered in the environment. After completing post-environment questionnaires, the participants are provided an opportunity to give verbal feedback about the experience and to note any observed problems with the interface or use of controllers, as well as their VR experience.

Study Duration: Phase 1 is expected to be completed in a period of 8 months from opening of enrollment to completion of data analysis. Phase 2 will require 12 months from opening of enrolment until data analysis.

Participant Duration: Phase 1 is completed in one visit to the NIH campus, Phase 2 may be completed in 1 or 2 visits to the NIH campus within the same week or consecutive weeks.

ELIGIBILITY:
* INCLUSION CRITERIA:

Male or female participant aged 18-75

Willingness to complete study procedures

Willing to provide feedback about VR experiences

Able to provide his/her own consent

EXCLUSION CRITERIA

Not fluent in English

Any impairment in visual functioning (e.g., 3-d depth perception, visual acuity, oculomotor control) not corrected with lenses

Eye pain or iritis

Susceptibility to photogenic seizures and/or diagnosis of seizure disorder

Inability to use hands to manipulate objects

Diagnosis of a neurological condition

Diagnosis of a sleep disorder

Current treatment for chronic physical pain, migraines, any diagnosis of a clinical condition associated with cognitive or physical fatigue (e.g. multiple sclerosis, chronic fatigue syndrome, etc.)

Any history of acquired brain injury

Current cold/flu symptoms

NINR employee/staff or subordinate, relative, and/or co-worker of NINR employee/staff or a study investigator.

For phase 2, participation in phase 1

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers from the Washington D.C. metropolitan area
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Phase 1: The total tally of the number of times a subject required research staff to explain how to use the controller, how to move or inspect objects, and/or how to move from one location to another location in the grocery store environment. | During study
  Phase 1: The outcome is the effectiveness of the grocery shopping training experience as indicated by the ability of healthy adults to perform all required shopping tasks in the immersive virtual reality environment.
Phase 2: The level of fatigue experienced after participating in a VR experience as measured by the Visual Analog Scale- Fatigue (VAS-F). | During study
  Phase 2: Self-reported change in cognitive fatigue.

SECONDARY OUTCOMES:
Obtain initial data pertaining to the environment's ability to create feelings of fatigue as intended. | During study
  Phase 1: secondary outcomes include: eye strain, level of presence in the virtual experience, cognitive load, and processing speed and working memory.
Identify performance and potential eye tracking measures that objectively identify fatigability. | During study
  Phase 2: Secondary outcomes include: ocular and physical symptoms pre- andpost shopping, evaluation of 1) shopping performance, 2) relationship between personality and subjective and objective fatigue susceptibility, 3) relationship between transient mood and trait fatigue and subjective and objective fatigue susceptibility, 4) relationship among subjective and objective fatigue measures, 5) relationships between individual characteristics and cognitive performance, fatigue, and workload.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Brennan, Ph.D., Principal Investigator — National Institute of Nursing Research (NINR)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Holdnack JA, Brennan PF. Usability and Effectiveness of Immersive Virtual Grocery Shopping for Assessing Cognitive Fatigue in Healthy Controls: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Aug 4;10(8):e28073. doi: 10.2196/28073. PMID 34346898
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001744-NR.html